CLINICAL TRIAL: NCT04050202
Title: Attachment and Biobehavioral Catch-up for Depression Intervention
Brief Title: Attachment and Biobehavioral Catch-up for Depression
Acronym: ABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A130886; K23MH113709 (NIH)
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Results first posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Depressive Symptoms; Anxiety Symptoms
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — abacavir; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABC (Experimental): ABC delivers therapy through 10, home-based, in-person sessions led by a trained professional. Treatment content is based on attachment theory and an understanding of children's stress neurobiology. Components aim to improve parental sensitivity, nurturance, and responsivity, as well as children's biological and behavioral reactivity through dyadic interactions between parents and children.
  Interventions: Behavioral: Attachment and Biobehavioral Catch-up (ABC) Intervention

INTERVENTIONS:
Behavioral: Attachment and Biobehavioral Catch-up (ABC) Intervention — ABC is a 10 session, home-based, dyadic therapy that is delivered by a trained professional. The sessions focus on improving the parent-child relationship and children's biological and behavioral responses to stress.
  Other Names: ABC

SUMMARY:
The overarching goal is to pilot the Attachment and Biobehavioral Catch-up (ABC) intervention for mothers with heightened depressive symptom and their children with heightened internalizing symptoms.

DETAILED DESCRIPTION:
Exposure to maternal depressive symptoms increases children's risk for developing anxiety and depressive symptoms ("internalizing symptoms"). Maternal depressive symptoms and children's internalizing symptoms may be reciprocally related over time. Optimal interventions for children's internalizing symptoms may involve treatment components for mothers, children, and the maternal-child relationship. The Attachment and Biobehavioral Catch-up (ABC) intervention is a empirically-supported, family-based treatment program that has been shown to be beneficial for children in varied high-risk family environments, but has yet to be tested among mothers and children recruited on the basis of heightened depressive and internalizing symptoms, respectively. The overarching goal is to examine the acceptability, feasibility, and preliminary effects of the ABC program on a sample of mother-child dyads (n = 20) with heightened depressive and internalizing symptoms. Our specific aims are:

1. To evaluate the feasibility and acceptability of ABC for mothers with depressive symptoms and their offspring with internalizing symptoms
2. To explore whether children who receive ABC show improvement in internalizing symptoms from pre- to post-intervention
3. To explore whether mothers who receive ABC show improvement in depressive symptoms from pre- to post-intervention
4. To explore whether parents and children who receive ABC show more adaptive physiological responses to stress from pre- to post-intervention

ELIGIBILITY:
Inclusion Criteria:

1. Mothers between 18 and 50 years of age with heightened depressive symptoms as determined by a score of 16 or higher on the Center for Epidemiologic Studies Depression Scale-Revised (CESD-R)
2. Biological children (of mothers described above) between 2 and 4 years old with heightened internalizing symptoms as determined by a T-score of 60 or higher on the Childhood Behavior Checklist (CBCL)

Exclusion Criteria:

* Self-reported history of psychosis or active suicidality as defined by self-report of a specific suicide plan or recent attempt
* Current pregnancy
* Child diagnosis of autism
* Pacemaker implant, cardiac problems, cardiac medication

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Roubinov, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between August 2020 and March 2021. Recruitment occurred online.
Pre-assignment Details: The numbers of enrolled participants reflect the total number of mothers and children. There were 21 dyads enrolled in the study reflecting 21 mothers and their 21 offspring (42 total participants).
Groups:
- Attachment and Biobehavioral Catch-up (ABC): ABC delivers therapy through 10 weekly sessions that are led by a trained professional ("parent coach"). Treatment content is based on attachment theory and an understanding of children's stress neurobiology. Components aim to improve parental sensitivity, nurturance, and responsivity. Parents are supported to improve the quality of their interactions with their children through frequent "in-the-moment" comments that are provided to them by the parent coach. All comments are positive initially; these comments highlight adaptive behaviors the parent is engaging in and the positive effect that they have on their children. Once rapport is established, the parent coach begins to offer suggested modifications or behaviors the parent may want to discontinue as they are likely to be dysregulating for the child.
Period: Overall Study
Arm/Group | Attachment and Biobehavioral Catch-up (ABC)
Started | 42 (There were 21 dyads who started the study reflecting 21 mothers and their 21 offspring (42 total participants).)
Completed | 40 (There were 20 dyads who started the study reflecting 20 mothers and their 20 offspring (40 total participants).)
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- Attachment and Biobehavioral Catch-up (ABC): ABC delivers therapy through 10 sessions led by a trained professional ("parent coach"). Treatment content is based on principles of attachment theory and an understanding of children's stress neurobiology. Each session is structured with content that aims to improve parental sensitivity, nurturance, and responsivity. Parents are provided with ongoing feedback ("in the moment" comments from the parent coach) that reinforces adaptive parenting behaviors and helps gently adapt non-adaptive or negative parenting behaviors.
Arm/Group | Attachment and Biobehavioral Catch-up (ABC)
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants] — There were 21 mothers between the age of 18 and 65. All offspring of these mothers were under the age of 18.
  Participants
    <=18 years | 21
    Between 18 and 65 years | 21
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: There were 21 mothers and 21 offspring. Age is reported separately for each. This sums to 42 total participants.
  years
    Maternal age: number analyzed (Participants) | 21
    Maternal age | 36.45 (4.05)
    Child age: number analyzed (Participants) | 21
    Child age | 2.82 (0.63)
Sex: Female, Male [Count of Participants; unit: Participants] — There were 21 mothers, all of whom were female. Of the 21 offspring, 3 were female and 18 were male. This sums to 24 female participants and 18 male participants. Population: There were 21 mothers and 21 offspring. Mothers and offspring data are reported separately, but sum to the overall number of baseline participants.
  Participants
    Mother: number analyzed (Participants) | 21
    Mother: Female | 21
    Mother: Male | 0
    Offspring: number analyzed (Participants) | 21
    Offspring: Female | 3
    Offspring: Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Maternal race and child race were collected separately. There were 21 mothers and 21 children, summing to the total of 42 participants.
  Participants
    Maternal race: number analyzed (Participants) | 21
    Maternal race: American Indian or Alaska Native | 0
    Maternal race: Asian | 7
    Maternal race: Native Hawaiian or Other Pacific Islander | 0
    Maternal race: Black or African American | 1
    Maternal race: White | 12
    Maternal race: More than one race | 0
    Maternal race: Unknown or Not Reported | 1
    Child race: number analyzed (Participants) | 21
    Child race: American Indian or Alaska Native | 0
    Child race: Asian | 2
    Child race: Native Hawaiian or Other Pacific Islander | 0
    Child race: Black or African American | 0
    Child race: White | 14
    Child race: More than one race | 5
    Child race: Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42
Center for Epidemiologic Studies Depression Scale (CES-D) [Mean (Standard Deviation); unit: units on a scale] — The CES-D is a validated self-report measure of depressive symptoms. Scores range from 0 to 60 with higher scores indicating more severe symptoms. Population: The CES-D is an adult measure of depressive symptoms. This information was only collected from the sample of mothers (n = 21).
  units on a scale
    number analyzed (Participants) | 21
    (all) | 26.57 (7.99)
Internalizing subscale of the Child Behavior Checklist (CBCL) [Mean (Standard Deviation); unit: units on a scale] — The internalizing subscale of the CBCL is a validated measure of emotional withdrawal, reactivity, sadness, anxiety, and other symptoms completed by mothers about their children. Scores range from 0 to 72 with higher scores indicating more severe symptoms. Population: The internalizing subscale measures child symptoms. It was only completed by mothers about the n = 21 children who participated in the study.
  units on a scale
    number analyzed (Participants) | 21
    (all) | 16.95 (9.56)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Internalizing Subscale Score of the Child Behavior Checklist (CBCL) at Week 10 (Value at Baseline Minus Value at Post Intervention (Week 10))
Description: The internalizing subscale of the CBCL is a validated measure of emotional withdrawal, reactivity, sadness, anxiety, and other symptoms completed by mothers about their children. Scores range from 0 to 72 with higher scores indicating more severe symptoms.
Time Frame: Change in score from baseline at post-intervention (week 10).
Population: Outcome data was completed by mothers for 20 children.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Attachment and Biobehavioral Catch-up (ABC): ABC is a 10 session intervention that aims to improve parental sensitivity, nurturance, and responsivity.
Arm/Group | Attachment and Biobehavioral Catch-up (ABC)
Number analyzed (Participants) | 20
units on a scale | 8.5 (6.09)
Statistical Analysis 1: Comparison: Attachment and Biobehavioral Catch-up (ABC); Test type: Other; p < 0.01, t-test, 2 sided; Mean Difference (Net) = 8.45 — The post-intervention score is subtracted from the baseline score

2. Primary Outcome: Change From Baseline in Center for Epidemiologic Studies-Depression Scale (CES-D) at Week 10 (Value at Baseline Minus Value at Post Intervention (Week 10))
Description: The CES-D is a validated self-report instrument of depressive symptoms. Scores range from 0 to 60 with higher values indicating more severe symptoms.
Time Frame: Change in score from baseline at post-intervention (week 10)
Population: Outcome data was completed by 20 mothers.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attachment and Biobehavioral Catch-up (ABC)
Number analyzed (Participants) | 20
units on a scale | 12.6 (7.73)
Statistical Analysis 1: Comparison: Attachment and Biobehavioral Catch-up (ABC); Test type: Other; p < 0.01, t-test, 2 sided; Mean Difference (Net) = 13.97 — The post-intervention score is subtracted from the baseline score

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a 1 year period.
Groups:
- Attachment and Biobehavioral Catch-up (ABC): ABC delivers therapy through 10, home-based, in-person sessions led by a trained professional. Treatment content is based on attachment theory and an understanding of children's stress neurobiology. Components aim to improve parental sensitivity, nurturance, and responsivity, as well as children's biological and behavioral reactivity through dyadic interactions between parents and children.
  Attachment and Biobehavioral Catch-up (ABC) Intervention: ABC is a 10 session, home-based, dyadic therapy that is delivered by a trained professional. The sessions focus on improving the parent-child relationship and children's biological and behavioral responses to stress.
Arm/Group | Attachment and Biobehavioral Catch-up (ABC)
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

LIMITATIONS AND CAVEATS:
Onset of the COVID-19 pandemic during the middle of the study. Some families completed the intervention in person and other families completed it virtually or a mix of in-person and virtual visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT04050202/Prot_SAP_000.pdf